CLINICAL TRIAL: NCT02792244
Title: First Time Mothers and Anal Incontinence Six Years Postpartum
Acronym: FiTMAI6
Status: Completed | Type: Observational
Sponsor: Ostfold Hospital Trust (Other)
Collaborators: St.Olavs Hospital, Trondheim University Hospital, Norway (Unknown); Norwegian University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hege Hølmo Johannessen, Post Doctor, Ostfold Hospital Trust
Other Study IDs: AB3299
Record Dates: First submitted 2016-06-02; First posted 2016-06-07 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Fecal Incontinence; Urinary Incontinence; Quality of Life
MeSH Terms: conditions — Fecal Incontinence; Urinary Incontinence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Previous studies show that incontinence is relatively common during pregnancy and after delivery. Experiencing incontinence during pregnancy or in the first year after delivery increases the risk of long term incontinence. There is scarce documentation of the long term prevalence of anal incontinence (AI) in Norway. This study aims to explore prevalence and risk factors for incontinence approximately six years after delivery among the 1718 who participated in two previous studies exploring the prevalence and predictors of anal incontinence in late pregnancy and during the first year after first delivery, and the effect of pelvic floor muscle exercises as treatment for anal incontinence after delivery. Increased awareness and knowledge about risk factors and long term prevalence of anal incontinence among health professionals as well as pregnant and parous women may give indications about which women to target for preventative measures to reduce the risk of new onset of postpartum AI during pregnancy and after delivery. Further, increased knowledge may aid in planning individualized follow-up during pregnancy and the first year as well as in the long term among women with existing AI symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Participants in previous studies

Exclusion Criteria:

* Women not participating in previous studies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parous women participating in two previous studies (1. primiparae delivering their first child between May 2009 and December2010 and 2. women with anal incontinence postpartum)
Sampling Method: Non-Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Anal incontinence | Anal incontinence six years postpartum
  St. Mark's score measuring frequency and severity of anal incontinence

SECONDARY OUTCOMES:
Urinary incontinence | urinary incontinence six years postpartum
  ICI-Q UI SF measuring frequency and severity of urinary incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Hege H Johannessen, PhD, Principal Investigator — Ostfold Hospital Trust

IPD SHARING:
Plan to Share IPD: No